CLINICAL TRIAL: NCT01463345
Title: Blood Conservation in Cardiac Surgery
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: PI left and closed study at Hackensack went to RUTGERS
Sponsor: Hackensack Meridian Health (Other)
Collaborators: Rutgers, The State University of New Jersey (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Pro00001949
Record Dates: First submitted 2011-10-27; First posted 2011-11-01 (Estimated); Last update posted 2018-07-24 (Actual); Status verified 2018-07

CONDITIONS: Transfusion Reactions; Post Cardiac Surgery
Keywords: Blood conservation; Transfusion; Hemoglobin trigger; Transfusion trigger; Cardiac surgery; Transfusion triggers post cardiac surgery
MeSH Terms: conditions — Transfusion Reaction | interventions — Blood Transfusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Conservative Transfusion Arm (Experimental): Subjects in the conservative transfusion arm will receive transfusion only when their hemoglobin levels reach 7.5 g/dl.
  Interventions: Other: Blood transfusion
- Liberal Transfusion Arm (Active Comparator): Subjects in the liberal transfusion arm will receive transfusion only when their hemoglobin levels reach 9.0 g/dl.
  Interventions: Other: Blood transfusion

INTERVENTIONS:
Other: Blood transfusion — Conservative transfusion arm: Subjects randomized to the conservative transfusion arm will receive transfusions of PRBCs post-surgery only when their Hgb level measures < 7.5 g/dl. Blood products should be given to maintain Hgb levels >7.5 g/dl.
  Arms: Conservative Transfusion Arm
Other: Blood transfusion — Liberal transfusion arm: Subjects randomized to the liberal transfusion arm will receive transfusions of PRBCs post-surgery only when their Hgb level measures < 9.0 g/dl. Blood products should be given to maintain Hgb levels > 9.0 g/dl.
  Arms: Liberal Transfusion Arm

SUMMARY:
The objective of the study is to examine the safety of two different hemoglobin (Hgb)-based transfusion triggers in patients post cardiac surgery.

DETAILED DESCRIPTION:
Nearly 20% of blood transfusions in the United States are given to in patients undergoing cardiac surgery. Despite the many blood conservation techniques that are available, safe, and efficacious for patients, many of these operations continue to be associated with significant amounts of blood usage. We believe that transfusion protocols which employ specific guidelines for transfusion can decrease blood product usage and improve outcomes for patients undergoing cardiac surgery. Our goal is to demonstrate that a carefully chosen trigger can achieve better outcomes.

Our hypothesis is that a transfusion trigger of Hgb 7.5 g/dl will lead to decreased utilization of blood transfusions and will have many positive effects on the patients post cardiac surgery in addition to substantial cost savings. We will use an evidence based approach to observe the relative safety of a conservative transfusion trigger (7.5 g/dl) as compared to a more liberal trigger (9.0 g/dl). We will also study the effect of blood conservation on the incidence of transfusion-related complications such as transfusion related lung injury (TRALI) and infectious complications as well as length of hospital stay, cost and ventilator time.

ELIGIBILITY:
Inclusion Criteria:

Subjects who meet all of the following criteria will be considered for inclusion in this study:

1. Subjects scheduled to undergo any of the following cardiac surgeries as part of their routine medical care:

   * CABG
   * AVR
   * MVR
   * MV Repair
   * CABG/AVR
   * CABG/MVR
   * CABG/MV Repair
   * Thoracic Aneurysm Repair ± any concomitant cardiac procedure (valve, CABG, etc.)
2. Subjects must be > 18 years of age
3. No prior history of cardiac surgery.
4. Able and willing to give informed consent

Exclusion Criteria:

Subjects who meet any of the following criteria will be excluded from participation in this study:

1. Prior history of cardiac surgery
2. Patients who do not have sufficient time prior to surgery to give proper informed consent (i.e.: immediate, emergency surgery)
3. Patients who are younger than 18 years of age
4. Prior history of

   * bleeding disorders
   * symptomatic anemia (i.e. persistent tachycardia, orthostatic hypotension, persistent pressor requirement)
   * hereditary/acquired coagulopathy
   * platelet defects (e.g.: disseminated intravascular coagulation (DIC), hemophilia, Henoch-Schönlein purpura, hereditary hemorrhagic telangiectasia, thrombocytopenia (ITP, TTP), thrombophilia, Von Willebrand's disease)
5. History of leukemia or any other blood related malignancy
6. History of liver failure
7. Current, or history of, pre-existing medical condition other than current cardiac condition, which in the opinion of the investigator, would place the subject at risk or have the potential to confound interpretation of the study results
8. Participation in another clinical trial
9. Lack of capacity to give informed consent.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-11; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Safety of the lower hemoglobin transfusion trigger of 7.5 g/dl against the higher hemoglobin transfusion trigger of 9.0 g/dl. | The assessment will last untill day 4 post surgery
  This outcome measure is a simultaneous assessment of the multiple end points duration of pressor use, symptomatic anemia, anemia-associated hypotension within 48 hours post surgery and Hgb recovery by day 4 post-surgery.

SECONDARY OUTCOMES:
Rate of incidence of transfusion related complications between the two randomizations arms. | This will be compared during the hospital stay, untill 30 days after discharge.
  The comparison will be based on a composite end point consisting of transfusion related lung injury (TRALI) that is ARDS, ventilator time>24 hours, pneumonia; stroke (permanent/transient); MI and renal failure.

CONTACTS AND LOCATIONS:
Overall Officials: Leonard Lee, M.D., Principal Investigator — Dr Lee is leaving Hackensack University Medical Center on June 30th, 2012. Effective July 1st, 2012 he will assume his new role as the Chief of Cardiothoracic Surgery Division at the University OF Medicine & Dentistry OFNew Jersey-Robert Wood Johnson
Locations (1):
- Hackensack University Medical Center, Hackensack, New Jersey, United States